CLINICAL TRIAL: NCT05587283
Title: Phase 1 Single-Centre, Double-Blind, Randomized, Placebo-Controlled, Multiple Ascending Dose Clinical Trial to Evaluate the Safety, Tolerability and Acceptability of Intravaginal Administration of LABTHERA-001 Capsules in Healthy Female Volunteers
Brief Title: Safety, Tolerability, and Acceptability Study of Intravaginal Administration of LABTHERA-001 Capsules in Healthy Women
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AtoGen Co. Ltd (Industry)
Collaborators: ATOGEN AUSTRALIA PTY LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: LT-001
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-10

CONDITIONS: Bacterial Vaginosis; Vaginal Disease; Bacterial Infections; Vaginitis; Infection, Bacterial
Keywords: LBP
MeSH Terms: conditions — Vaginosis, Bacterial; Vaginal Diseases; Bacterial Infections; Vaginitis | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Eight participants will be randomized to be allocated into either a treatment group or a placebo control group (3:1 ratio) for each cohort. There will be three ascending dose cohorts. For the first two doses, the next dose cohorts will begin enrollment only after the safety data review meets a satisfactory evaluation by the safety review committee.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Low dose LABTHERA-001 capsule (Experimental): Low dose LABTHERA-001 capsule (0.2 x 10^9 CFU), administered intravaginally once a day for 7 consecutive days.
  Interventions: Drug: Experimental: Low dose LABTHERA-001 capsule
- Medium dose LABTHERA-001 capsule (Experimental): Medium dose LABTHERA-001 capsule (1 x 10^9 CFU), administered intravaginally once a day for 7 consecutive days.
  Interventions: Drug: Experimental: Medium dose LABTHERA-001 capsule
- High dose LABTHERA-001 capsule (Experimental): High dose LABTHERA-001 capsule (5 x 10^9 CFU), administered intravaginally once a day for 7 consecutive days.
  Interventions: Drug: Experimental: High dose LABTHERA-001 capsule
- Low dose Placebo capsule (Placebo Comparator): Low dose Placebo (excipients of the study drug) capsule administered intravaginally once a day for 7 consecutive days.
  Interventions: Other: Placebo Comparator: Low dose Placebo capsule
- Medium dose Placebo capsule (Placebo Comparator): Medium dose Placebo capsule (excipients of the study drug) administered intravaginally once a day for 7 consecutive days.
  Interventions: Other: Placebo Comparator: Medium dose Placebo capsule
- High dose Placebo capsule (Placebo Comparator): High dose Placebo capsule (excipients of the study drug) administered intravaginally once a day for 7 consecutive days.
  Interventions: Other: Placebo Comparator: High dose Placebo capsule

INTERVENTIONS:
Drug: Experimental: Low dose LABTHERA-001 capsule — Low dose LABTHERA-001 capsule, 0.2 x 10^9 CFU/capsule with excipients.
  Other Names: Lactobacillus Plantarum ATG-K2
  Arms: Low dose LABTHERA-001 capsule
Drug: Experimental: Medium dose LABTHERA-001 capsule — Medium dose LABTHERA-001 capsule, 1 x 10^9 CFU/capsule with excipients.
  Other Names: Lactobacillus Plantarum ATG-K2
  Arms: Medium dose LABTHERA-001 capsule
Drug: Experimental: High dose LABTHERA-001 capsule — High dose LABTHERA-001 capsule, 5 x 10^9 CFU/capsule with excipients.
  Other Names: Lactobacillus Plantarum ATG-K2
  Arms: High dose LABTHERA-001 capsule
Other: Placebo Comparator: Low dose Placebo capsule — Medium dose Placebo capsule, filled with excipients; Lactose, and magnesium stearate.
  Other Names: Control substance
  Arms: Low dose Placebo capsule
Other: Placebo Comparator: Medium dose Placebo capsule — Medium dose Placebo capsule, filled with excipients; Lactose, and magnesium stearate.
  Other Names: Control substance
  Arms: Medium dose Placebo capsule
Other: Placebo Comparator: High dose Placebo capsule — High dose Placebo capsule, filled with excipients; Lactose, and magnesium stearate.
  Other Names: Control substance
  Arms: High dose Placebo capsule

SUMMARY:
This is a phase 1, Single-Center, Double-Blind, Randomized, Placebo-Controlled, dose escalation, clinical trial enrolling 24 healthy participants. The main subject is to investigate the safety and tolerability of the LABTHERA-001 capsule and to explore the acceptability of the capsule.

DETAILED DESCRIPTION:
Bacterial vaginosis (BV) is the most common vaginal syndrome frequently found in women. BV is currently mainly treated with antibiotics. However, antibiotic administration can cause various side effects. And one of them is destroying the normal bacteria in the vagina, affecting the balance of the vaginal flora, increasing the likelihood of bacterial vaginosis recurrence, and causing drug resistance of bacteria. Therefore, the importance of fundamental treatment with the recovery of balance in normal vaginal flora is being recognized increasingly. The study drug for this trial, LABTHERA-001, has been derived from the bacteria Lactobacillus plantarum ATG-K2. Administration of the ATG-K2 strain will temporarily colonize the vagina to encourage a more normal microbiome.

The main goals of this study are 1. to determine whether LABTHERA-001 is safe and well tolerated in healthy adult women. And 2. to investigate the acceptability of the LABTHERA-001 capsule or matching placebo by completing a satisfaction evaluation questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy non-smoking woman aged 18 to 45 years old as of the date of written consent
2. Agrees to maintain her contraceptive method during the clinical trial if she has regular menstrual cycles (21-35 days) or has had amenorrhea for more than 12 weeks before the Screening Visit due to continued use of long-acting progestin or oral contraceptives.
3. Confirmed normal cervical screen test (CST) performed at the Screening Visit
4. Has had sexual experiences that included vaginal intercourse
5. Has experienced gynecological examinations previously
6. Agrees to discontinue the use of the following during the clinical trial period (Screening Visit to End of study visit or early termination visit):

   * products for vaginal insertion (e.g., tampons, menstrual cups, etc.)
   * Other vaginal products (e.g., contraceptive creams, vaginal cleaners, lubricants, etc.)
7. Agrees to be sexually abstinent from 72 hours before the Day 1 visit until the first study visit after final administration of IP (nominally the Day 9 visit).
8. Agrees to continue to use the following highly effective contraceptive methods during the clinical trial period and for at least 30 days after the final dose of study treatment, if woman of child-bearing potential (has experienced menarche and is not permanently sterile or postmenopausal):

   * Female: combined (estrogen and progestogen containing) hormonal/ contraception associated with inhibition of ovulation (oral or transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device (IUD; if inserted more than 12 weeks before the Screening visit), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner, sexual abstinence
   * Male partner: 'Vasectomy,' 'condom'
9. Able and willing to insert a hard capsule into her vagina
10. Able and willing to answer questions about her health status and sexual life
11. Able and willing to undergo vaginal and cervical examinations by the Investigator
12. Agrees and can comply with the planned clinical trial procedures after receiving a full explanation and voluntarily decides to participate and gives written informed consent

Exclusion Criteria:

1. Confirmed to have the following urogenital infections from the vaginal discharge test performed at the Screening Visit, or had the following diagnosed urogenital infections within three weeks before the Screening Visit, or has a history of clinically significant urogenital infections at the discretion of the Investigator:

   • Urinary tract infection, bacterial vaginosis, candida vaginitis, trichomonas vaginalis, Neisseria gonorrhoeae, chlamydia trachomatis, treponema pallidum, herpes simplex
2. History of recurrent genital herpes
3. Has the following diagnosed urogenital infections, or had two or more clinically significant urogenital infections within 24 weeks before the Screening Visit, at the discretion of the Investigator:

   • [Gonococcus, chlamydia trachomatis, syphilis treponema, trichomonas vaginitis, candida vaginitis, etc.]
4. Has vaginitis symptoms (abnormal vaginal discharge, itching, burning sensation, etc.) at Screening or pre-dose at the Day 1 visit, or between the Screening and Day 1 visits.
5. Is pregnant, lactating, within eight weeks of childbirth, or is planning pregnancy within 60 days of the last dose of IP.
6. Is menopausal, defined as being amenorrhoeic for at least 12 months without an alternative cause.
7. Has had an intrauterine device (IUD) inserted within 12 weeks before the Screening Visit
8. Underwent pelvic surgery within 12 weeks before the Screening Visit
9. Received cervical cryotherapy or cervical laser treatment within 12 weeks before the Screening Visit
10. Started to use long-acting hormonal contraceptives within 12 weeks before the Screening Visit [e.g., DMPA (depot formulation including medroxyprogesterone acetate)] (However, participants who have continuously used the contraceptive for more than 12 weeks can be enrolled at the discretion of the Investigator.)
11. Has a clinically significant medical history or current medical condition as assessed by the Investigator including but not limited to the cardiovascular system, respiratory system, kidney, endocrine system, hematology, digestive system, central nervous system, psychiatric disorder, or infectious disease, that may affect the safety evaluation of the investigational product or jeopardize the individual's involvement in the study. History of any cancer (including non-melanoma skin cancer) is exclusionary.
12. Positive test for SARS-CoV-2 (COVID-19) during the Screening period and pre-dose at the Day 1 visit (may be re-screened when eligible).
13. Positive diagnosis of human immunodeficiency virus (HIV), hepatitis B or C at the Screening Visit
14. Confirmed to have severe damage to the vaginal epithelium in the physical examination at the Screening Visit
15. Used immunosuppressants within four weeks before the Screening Visit
16. Used antibiotics or antifungals within three days before the Screening Visit (However, enrollment is possible if the individual agrees to a washout period equivalent to three times or more the half-life of the corresponding drugs as of the randomization date.)
17. History of hypersensitivity reactions to the components of the study drug or history of other serious drug hypersensitivity reactions, at the discretion of the Investigator
18. History of or current drug or alcohol abuse; or tests positive to urine drug screen or alcohol breath test at the Screening or Day 1 visits; or does not agree to abstain from alcohol 24 hours before each study visit and to consume no more than 10 standard drinks per week with no more than 4 standard drinks on any one day at any other time during their participation in the study. One standard drink contains 10 g alcohol. Urine drug screen may be repeated once only at the discretion of the Investigator.
19. Current tobacco smoker; or smoked more than one pack of cigarettes (or tobacco equivalent) per day for more than 10 years; or uses nicotine-replacement therapy (including vaping); or does not agree to abstain from using tobacco or nicotine-containing products during the study.
20. Received other investigational products within four weeks before the Screening Visit
21. Received COVID-19 vaccination or any other vaccination within 8 weeks before the first dose of IP, and/or is planning or scheduled to be vaccinated (including COVID-19 initial, second or booster dose) during the study period up to the final follow-up visit.
22. Judged by the Investigator to be unsuitable for participation in this clinical trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Number of AEs in participants throughout the study and their severity and relationship to the study product. | 35 days since the first dose administration
  Any incidence of adverse events will be evaluated for their severity and relationship to the study product. The number of AEs and other combined measurement results will be evaluated for the safety of the study product.
Changes in Clinical Laboratory Tests, Vital signs (body temperature, respiratory rate, heart rate, blood pressure), Gynaecological Examination, and Physical Examination. | Baseline and each follow-up visit upto 35 days since the first dose administration (Day 1)
  Day 1 pre-dose results will be used as the baseline values. Abnormalities in clinical laboratory parameters, gynaecological examination findings, and vital signs will be based on predefined normal ranges and will be tabulated by dose group showing participant counts and percentages.

SECONDARY OUTCOMES:
Acceptability evaluation | Visit 3 (Day 9)
  5-point Likert scale, 1 (strongly disagree), 2 (disagree), 3 (neither disagree or agree), 4 (agree), and 5 (strongly agree), in response to 7 statements at visit 3 (Day 9) to evaluate how acceptable participants found using the study product.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Argent, Dr., Principal Investigator — Scientia Clinical Research Ltd
Locations (1):
- Scientia Clinical Research, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mastromarino P, Vitali B, Mosca L. Bacterial vaginosis: a review on clinical trials with probiotics. New Microbiol. 2013 Jul;36(3):229-38. Epub 2013 Jun 30. PMID 23912864
- [Background] Kenyon C, Colebunders R, Crucitti T. The global epidemiology of bacterial vaginosis: a systematic review. Am J Obstet Gynecol. 2013 Dec;209(6):505-23. doi: 10.1016/j.ajog.2013.05.006. Epub 2013 May 6. PMID 23659989
- [Background] Workowski KA, Bachmann LH, Chan PA, Johnston CM, Muzny CA, Park I, Reno H, Zenilman JM, Bolan GA. Sexually Transmitted Infections Treatment Guidelines, 2021. MMWR Recomm Rep. 2021 Jul 23;70(4):1-187. doi: 10.15585/mmwr.rr7004a1. PMID 34292926
- [Background] Vicariotto F, Mogna L, Del Piano M. Effectiveness of the two microorganisms Lactobacillus fermentum LF15 and Lactobacillus plantarum LP01, formulated in slow-release vaginal tablets, in women affected by bacterial vaginosis: a pilot study. J Clin Gastroenterol. 2014 Nov-Dec;48 Suppl 1:S106-12. doi: 10.1097/MCG.0000000000000226. PMID 25291116
- [Background] De Seta F, Parazzini F, De Leo R, Banco R, Maso GP, De Santo D, Sartore A, Stabile G, Inglese S, Tonon M, Restaino S. Lactobacillus plantarum P17630 for preventing Candida vaginitis recurrence: a retrospective comparative study. Eur J Obstet Gynecol Reprod Biol. 2014 Nov;182:136-9. doi: 10.1016/j.ejogrb.2014.09.018. Epub 2014 Sep 17. PMID 25305660
- [Background] Strus M, Chmielarczyk A, Kochan P, Adamski P, Chelmicki Z, Chelmicki A, Palucha A, Heczko PB. Studies on the effects of probiotic Lactobacillus mixture given orally on vaginal and rectal colonization and on parameters of vaginal health in women with intermediate vaginal flora. Eur J Obstet Gynecol Reprod Biol. 2012 Aug;163(2):210-5. doi: 10.1016/j.ejogrb.2012.05.001. Epub 2012 Jun 19. PMID 22721635
- [Background] Hemalatha R, Mastromarino P, Ramalaxmi BA, Balakrishna NV, Sesikeran B. Effectiveness of vaginal tablets containing lactobacilli versus pH tablets on vaginal health and inflammatory cytokines: a randomized, double-blind study. Eur J Clin Microbiol Infect Dis. 2012 Nov;31(11):3097-105. doi: 10.1007/s10096-012-1671-1. Epub 2012 Jul 10. PMID 22777592